## #MoveUp Study New York State Psychiatric Institute/Columbia U 1051 Riverside Dr, New York NY 10032 646-774-6965

NYSPI IRB Approved 7574 12/14/2020 -> 11/12/2021

## AUTHORIZATION FOR THE RELEASE OF INFORMATION

| I | , herby authorize and give my | |
|---|---|---|
| permission | n to the <u>#MoveUp Study, New York Psychiatric I</u> | nstitute/Columbia University, |
| 1051 River | rside Dr, New York, New York 10032 to release/ | receive information limited to |
| the follow: | ring specific items: | |
| • Na | ame and contact information of study participant | |
| • Re | eason(s) for referral to treatment | |
| • Da | ate(s) of attendance at intake and/or treatment ses | sions |
| • Da | ate(s) of clinic/agency visits | |
| • Da | ate(s) of treatment received | |
| • De | escription of treatment received | |
| - | ne confidential information to be released or recei<br>gencies, or organizations: | ved only to/from the following |
| I permit th | nis confidential information to be released only fo | r the following reasons and |
| • Da | ata collection for the #MoveUp study | |
| • As | ssistance with linkage and referrals for treatment | |
| any time, e | prization to release confidential information may be except to the extent that action has already been to make the released without the execution of an add | aken; no further confidential |
| Date | of Permission | Signature of Participant |
| | | Signature of #MoveUp Staff |